CLINICAL TRIAL: NCT07060105
Title: Efficacy of Hypertonic Saline as a Treatment for Mild Traumatic Brain Injury in Pediatric Patients
Brief Title: Hypertonic Saline for Mild TBI in Pediatric Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lina Palomares, Clinical Research Coordinator, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 00004358
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Head Injury, Minor; Pediatric; Emergency Department Patient
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Saline (Experimental): The intervention group (n=37) will receive 5ml/kg of 3% hypertonic saline
  Interventions: Other: Hypertonic Saline ( 3% Sodium Chloride Saline)
- Normal Saline (Active Comparator): Control group (n=37) will receive 5ml/kg of 0.9% normal saline
  Interventions: Other: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Other: Hypertonic Saline ( 3% Sodium Chloride Saline) — The intervention group (n=37) will receive 5ml/kg of 3% hypertonic saline, and the control group (n=37) will receive 5ml/kg of 0.9% normal saline. There is a maximum volume of 500ml for both fluids.
  Arms: Hypertonic Saline
Other: Normal Saline (0.9% NaCl) — The intervention group (n=37) will receive 5ml/kg of 3% hypertonic saline, and the control group (n=37) will receive 5ml/kg of 0.9% normal saline. There is a maximum volume of 500ml for both fluids.
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to compare two different treatments (normal saline and hypertonic saline) for concussions to see if one makes more of a difference in symptoms that can occur following concussions.

DETAILED DESCRIPTION:
This randomized, double-blinded prospective study aims to determine the utility and efficacy of 3% hypertonic saline (HTS) to combat acute and long-term sequelae of TBI. We plan to enroll 74 participants, ages 8-17, who present to the pediatric Emergency Department with a mild TBI. The intervention group (n=37) will receive 5ml/kg of 3% hypertonic saline, and the control group (n=37) will receive 5ml/kg of 0.9% normal saline. There is a maximum volume of 500ml for both fluids. A standardized concussion inventory score will be used to assess the severity of symptoms pre-infusion, and post-infusion. Participants (or their parent/guardian) will be asked to complete two additional inventory scores one week and one month after the injury, of which they will be reimbursed for successful completion. Primary outcomes will be the efficacy of HTS in treating acute and chronic concussion symptomatology, and secondary outcomes will include unscheduled revisits to the ED.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-17
2. Blunt head injury within the past five days with any associated symptoms as outlined in the concussion inventory.
3. English or Spanish speaking.
4. Glasgow Coma Scale score of 13-15
5. Treating provider plans to use saline administration as part of patient's treatment plan

Exclusion Criteria:

1. Intracranial injury diagnosed by CT / MR Brain, though imaging is not a requirement for this study.
2. Possible or witnessed posttraumatic seizure
3. Developmental delay / intellectual disability
4. Underlying cardiac, pulmonary, and renal pathology in which fluid administration or hypertonic saline may potentially be harmful, based on attending provider judgement.
5. Suspected use of alcohol or illicit substances
6. Associated injuries requiring the use of narcotics for analgesia

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Concussion symptoms severity | One month
  A standardized concussion inventory score will be used to assess the severity of symptoms pre-infusion, and post-infusion. Participants (or their parent/guardian) will be asked to complete two additional inventory scores one week and one month after the injury, of which they will be reimbursed for successful completion. Primary outcomes will be the efficacy of HTS in treating acute and chronic concussion symptomatology.
Severity of concussion symptoms | One month
  A standardized concussion inventory score will be used to assess the severity of symptoms pre-infusion, and post-infusion. Participants (or their parent/guardian) will be asked to complete two additional inventory scores one week and one month after the injury, of which they will be reimbursed for successful completion. Primary outcomes will be the efficacy of HTS in treating acute and chronic concussion symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wilkinson, MD, MPH, Principal Investigator — The University of Texas at Austin
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to maintain participant confidentiality. Aggregate data requests will be reviewed.

REFERENCES:
- See also: Study information site — https://sites.utexas.edu/pem-research-lab/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT07060105/Prot_SAP_000.pdf